CLINICAL TRIAL: NCT06572202
Title: Effectiveness of Positive Psychological Intervention on Resilience Improvement in Nurses: A Randomised Controlled Trial
Brief Title: Effectiveness of Positive Psychological Intervention on Resilience Improvement in Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fitria Endah Janitra (Other)
Responsible Party: Sponsor-Investigator, Fitria Endah Janitra, Principal Investigator, Taipei Medical University
Organization: Taipei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FRESPP2024
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Nurses; Resilience, Psychological; Positive Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology Intervention (Experimental): The experimental group will receive multicomponent of positive psychology intervention with the specific domain related to resilience enhancement in nurses Ciarrochi et al. (2022). The program consists of five resilience domains/ six positive psychology virtues in fourteen sessions. Each session will take 60 minutes, two sessions per week. The program will last for six weeks, followed by posttest immediately after intervention, 3-months, 6-months, and one year follow up.
  Interventions: Behavioral: Positive Psychology Intervention
- Control group (No Intervention): The control group will not receive intervention

INTERVENTIONS:
Behavioral: Positive Psychology Intervention — The 14-session intervention program is designed to enhance various internal resiliency factors. It begins with an orientation to positive psychology and setting group guidelines. Cognitive resilience is developed through identifying personal and signature strengths, reappraising memories, and learning savoring techniques. Emotional resilience is strengthened by focusing on forgiveness, managing decision fatigue, and fostering positive communication. Spiritual resilience is cultivated through gratitude practices and exploring hope and optimism. Behavioral resilience is addressed by recognizing strengths in others and engaging in altruism. The final session integrates all these elements to promote lasting positive changes in engagement, relationships, meaning, and accomplishments. Mid-session feedback ensures the program's effectiveness and responsiveness to participants' needs.
  Arms: Positive Psychology Intervention

SUMMARY:
The nursing profession, comprising over 27.9 million individuals and representing 59% of the health sector, plays a critical role in frontline healthcare globally. However, nurses face significant workplace stress due to factors like high mortality rates and ethical dilemmas, which can negatively impact their mental health. Resilience has emerged as a crucial concept in mitigating workplace stress and protecting nurses' psychological well-being. Studies show a negative correlation between stress and resilience, with higher resilience linked to better psychological outcomes and lower rates of burnout. Resilience, a dynamic process of positive adaptation to stress, can be enhanced through interventions like positive psychology, which focuses on developing traits such as perseverance, interpersonal skills, and emotional stability. These interventions have been shown to reduce burnout, improve job satisfaction, and potentially enhance patient care, making them vital in addressing the unique challenges nurses face.

Gap of Knowledge:

Although existing research has demonstrated the effectiveness of positive psychology interventions in reducing depression, anxiety, burnout, and stress among healthcare workers, including nurses, there is a need for more targeted randomized controlled trials (RCTs) that specifically address the unique stressors and work environments of nurses. Furthermore, the long-term effects of these interventions on nurses' resilience, stress, burnout, and job satisfaction require further exploration through well-designed RCTs.

Research Aims and Hypothesis:

The present study aims to

1. evaluate whether a positive psychology intervention, based on evidence-based activities from several positive psychology theories, can improve resilience in nurses, and
2. assess whether this intervention can also enhance stress levels, reduce burnout, and improve job satisfaction among nurses.

The hypotheses are:

1. the positive psychology intervention will improve nurses' resilience;
2. the intervention will positively impact stress, burnout, and job satisfaction; and
3. it will be more effective for nurses with low resilience in improving these outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. registered nurses working in clinical settings
2. minimum of one year of work experience as a nurse
3. availability to participate in the intervention and follow-up assessments.

Exclusion Criteria:

1. Recent exposure to severe illness, trauma, or major life events in the past three months,
2. having suffered a major traumatic event in the past 6 months,
3. currently undergoing other forms of psychological treatment or counseling.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2025-03-09 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
Resilience | pre-test, immediately after intervention, 3 months follow-up, 6 months follow-up, 12 month follow-up
  Resilience will be measure with the Connor Davidson Resilience Scale (CD-RISC). The CD-RISC was developed in the United States to measure individuals' ability to cope effectively when faced with adversity (Connor & Davidson, 2003). The revised scale includes 25 items and three dimensions (tenacity, strength, and optimism). Each item is rated on a Likert-type scale ranging from 0 (not at all) to 4 (almost always). The Cronbach's alpha value for the CDRISC 25 has been reported to be 0.91 in a study on a sample of nurses (Arias González et al., 2015).

SECONDARY OUTCOMES:
Stress | pre-test, immediately after intervention, 3 months follow-up, 6 months follow-up, 12 month follow-up
  Stress will be measured by the Perceived Stress Scale (PSS). The PSS-10 is a 10-item questionnaire that is widely used to assess stress levels in young people and adults aged 12 and above. The Cronbach's alpha value for the Perceived Stress Scale (PSS-10) in nurses has been reported to be 0.93 in a study in South Africa (Engelbrecht, 2022).
Anxiety | pre-test, immediately after intervention, 3 months follow-up, 6 months follow-up, 12 month follow-up
  Anxiety will be measured using the Generalized Anxiety Disorder 7 (GAD-7) scale. The GAD-7 is a brief, seven-item self-report questionnaire designed to identify probable cases of generalized anxiety disorder and to measure the severity of the symptoms. The Cronbach's alpha for the GAD-7 has been reported to be 0.92 in a study by Spitzer et al. (2006).
Depression | pre-test, immediately after intervention, 3 months follow-up, 6 months follow-up, 12 month follow-up
  Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a nine-item self-report tool that is used to screen for the presence and severity of depression. Each item is scored from 0 to 3, providing a total score ranging from 0 to 27, with higher scores indicating greater severity of depressive symptoms. The Cronbach's alpha for the PHQ-9 has been reported to be 0.89 in a study by Kroenke et al. (2001).
Burnout | pre-test, immediately after intervention, 3 months follow-up, 6 months follow-up, 12 month follow-up
  Burnout will be measure with The Maslach Burnout Inventory (MBI). MBI is a psychological assessment instrument that measures burnout as a continuum on three different dimensions: Emotional Exhaustion, Depersonalization, and reduced Personal Accomplishment. The MBI is considered the "gold standard" for measuring burnout. The Cronbach's alpha value for the Maslach Burnout Inventory (MBI) in nurses has been reported to range from 0.70 to 0.90, indicating good internal consistency and reliability (Trigo et al., 2018).
Work performance | pre-test, immediately after intervention, 3 months follow-up, 6 months follow-up, 12 month follow-up
  Work performance will be measured by the Individual Work Performance Questionnaire (IWPQ). The IWPQ assesses individual work performance across three dimensions: task performance, contextual performance, and counterproductive work behavior. This questionnaire includes items that evaluate how well nurses plan and execute their work, their willingness to help colleagues and take on additional responsibilities, and their ability to avoid counterproductive behaviors. The IWPQ is known for its reliability, with Cronbach's alpha values typically ranging from 0.70 to 0.85 across different dimensions, making it a dependable tool for measuring work performance.
Physical health | pre-test, immediately after intervention, 3 months follow-up, 6 months follow-up, 12 month follow-up
  To measure physical health outcomes, blood pressure will be assessed. Blood pressure will be assessed using automated blood pressure monitors, which provide reliable and easy-to-use measurements of both systolic and diastolic pressures.

CONTACTS AND LOCATIONS:
Overall Officials: Fitria Endah Janitra, Principal Investigator — Universitas Islam Sultan Agung
Locations (1):
- Sultan Agung Islamic Teaching Hospital, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silva Ddos S, Tavares NV, Alexandre AR, Freitas DA, Breda MZ, Albuquerque MC, Melo VL. [Depression and suicide risk among nursing professionals: an integrative review]. Rev Esc Enferm USP. 2015 Dec;49(6):1027-36. doi: 10.1590/S0080-623420150000600020. Portuguese. PMID 27419688
- [Result] Aqtam I, Ayed A, Toqan D, Salameh B, Abd Elhay ES, Zaben K, Mohammad Shouli M. The Relationship Between Stress and Resilience of Nurses in Intensive Care Units During the COVID-19 Pandemic. Inquiry. 2023 Jan-Dec;60:469580231179876. doi: 10.1177/00469580231179876. PMID 37278278
- [Result] Mealer M, Jones J, Newman J, McFann KK, Rothbaum B, Moss M. The presence of resilience is associated with a healthier psychological profile in intensive care unit (ICU) nurses: results of a national survey. Int J Nurs Stud. 2012 Mar;49(3):292-9. doi: 10.1016/j.ijnurstu.2011.09.015. Epub 2011 Oct 5. PMID 21974793
- [Result] Janitra FE, Jen HJ, Chu H, Chen R, Pien LC, Liu D, Lai YJ, Banda KJ, Lee TY, Lin HC, Chang CY, Chou KR. Global prevalence of low resilience among the general population and health professionals during the COVID-19 pandemic: A meta-analysis. J Affect Disord. 2023 Jul 1;332:29-46. doi: 10.1016/j.jad.2023.03.077. Epub 2023 Mar 31. PMID 37004902